CLINICAL TRIAL: NCT00200239
Title: Provision of Breakfast Food in Behavioral Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2047-05
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2007-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

ARMS (2):
- 1 (Experimental): Behavioral: eating breakfast from portioned and unportioned foods
  Interventions: Behavioral: Eating breakfast with portion and unportioned foods
- 2 (Experimental): Behavioral: eating breakfast with portioned and unportioned foods
  Interventions: Behavioral: Eating breakfast with portion and unportioned foods

INTERVENTIONS:
Behavioral: Eating breakfast with portion and unportioned foods — Behavioral: eating breakfast with portion and unportioned foods

SUMMARY:
A contributing factor to the rising prevalence of obesity may be increased portion sizes. However, the effect of portion size has not been studied independent of the effect of quantity of food in the context of a behavioral weight loss program. Providing pre-portioned single servings of food may make it easier to reduce caloric and dietary fat intake improving weight loss. In addition, breakfast skipping is associated with obesity and breakfast consumption is associated with weight loss success. Therefore, the objective of the proposed study is to investigate the effect of portion size on consumption of provided breakfast foods in the context of a behavioral weight loss program. Participants will be randomized to 1 of 2 standard 12-week behavioral obesity interventions. The first intervention, serving as a control, will provide participants with breakfast foods in non-portioned containers (Standard). A second intervention will provide participants with the same type and quantity of breakfast foods but they will be provided in pre-portioned single servings (Portion). Dependent variables include the number of calories consumed from the provided foods as well as overall caloric and fat consumption. If the provision of food in pre-portioned servings is effective at decreasing intake, future directions include conducting longer interventions to improve long-term weight loss outcomes in standard behavioral interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 21 and 65 years. Older adults may have more medical co-morbidities and may require greater medical supervision.
2. Body mass index (BMI) between 25 and 40 kg/m2. Based upon the Evidence Report (National Heart, Lung, and Blood Institute [NHLBI], 1998), weight loss is recommended for individuals with a BMI > 25. However, individuals with a BMI of > 40 have more medical co-morbidities and require greater medical supervision.
3. Average current consumption of breakfast on four days or fewer.

Exclusion Criteria:

1. Report allergies to any of the foods provided in the treatment or report lactose intolerance due to the high lactose content of some of the foods provided.
2. Report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q) (Thomas, Reading, & Shephard, 1992). Individuals endorsing joint problems, prescription medication usage, or other medical conditions that could limit exercise will be required to obtain written physician consent to participate.
3. Report major psychiatric diseases or organic brain syndromes.
4. Are currently participating in a weight loss program and/or taking weight loss medication or lost > 5% of body weight during the past 6 months.
5. Intend to move to another city within the time frame of the investigation or will be out of town and unavailable for meetings for more than one week during the treatment program.
6. Are pregnant, lactating, less than 6 months post-partum, or plan to become pregnant during the time frame of the investigation.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2005-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Intake of breakfast foods | 8 weeks

SECONDARY OUTCOMES:
Weight loss | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, PhD, Principal Investigator — University of Tennessee
Locations (1):
- The Weight Control and Diabetes Research Center, Providence, Rhode Island, United States